CLINICAL TRIAL: NCT07074184
Title: Radiofrequency Intervention in Musculoskeletal Pathologies Post COVID-19
Brief Title: Radiofrequency Intervention in Post-COVID-19 Patients With Musculoskeletal Sequelae
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinica Gema Leon (Other)
Responsible Party: Principal Investigator, GEMA LEÓN BRAVO, Investigador Principal, Clinica Gema Leon
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ART-GLB-RF-MUSC-COVID
Record Dates: First submitted 2025-07-16; First posted 2025-07-20 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Covid19; Musculoskeletal Injury
Keywords: COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Musculoskeletal Manipulations

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo group (Placebo Comparator): Placebo Group: Patient receiving treatment with radiofrequency turned off
  Interventions: Other: Turn off radiofrequency 448khz
- Treatment group (Experimental): Experimental Mixed Group: Patient receiving treatment with manual therapy and radiofrequency;
  Interventions: Other: Radiofrequency 448khz with manual therapy
- Conventional group (Active Comparator): Convencional Manual Group: Patient receiving treatment with manual therapy
  Interventions: Other: Manual therapy

INTERVENTIONS:
Other: Radiofrequency 448khz with manual therapy — The intervention in consisted of a total of 12 sessions (twice a week) of treatment. The set duration for each session was 45 minutes, except for those sessions where variable measurements were required, which lasted 60 minutes. Radiofrequency 448 Hz was administered to the affected area in two phases, depending on the electrode applied: 5 minutes of capacitive electrode and 25 minutes of resistive electrode. In addition, a specific joint physical therapy manual therapy treatment was also performed, in which pumping techniques were performed after the radiofrequency treatment.
  Arms: Treatment group
Other: Turn off radiofrequency 448khz — Radiofrequency 448 Hz was administered to the affected area in two phases, depending on the electrode applied: 10 minutes of capacitive electrode and 35 minutes of resistive electrode, both with the machine turned off.
  Arms: Placebo group
Other: Manual therapy — Articulatory pumping techniques were applied towards the painful position with the aim of reducing it.
  Arms: Conventional group

SUMMARY:
The sequelae that occur in post-COVID-19 patients are multiple and, at a therapeutic level, these represent a new challenge within the general context of the pandemic that the world is suffering.

The virus has managed to end thousands of lives today and many other cases are being charged as directly responsible for a multiplicity of multisystem damages that need to be diagnosed and treated. Among the most relevant, are those that can affect to levels musculoskeletal in patients without previous pathologies, and in patients at risk who already had a pathology prior to infection.

On the other hand, signs and symptoms have been observed characteristic in the organ systems described above in post-contagion patients, directly associated with sequelae SARV-CoV2. The radiofrequency (RF) of electromagnetic waves represents a technology of proven efficacy and safety in multiple fields of both human and veterinary medicine. These include neurological and pneumological pathologies, and very especially those that affect the locomotor system. In therapeutics there are different RF modalities depending on the modality, polarity, type of signal and frequency, which in turn translate into different therapeutic profiles, clinical indications, efficacy and safety.

Among the RF technologies most used today and that have a greater scientific background, is the one known as Resistive Capacitive Monopolar Radio Frequency at 448 kHz (INDIBA®). This study aims to assess the efficacy and safety of RFMCR in the treatment of musculoskeletal sequelae in patients presenting this type of pathologies that appear after contagion by COVID-19. Through this non-invasive technique, the investigators want to show that RF can help the physical rehabilitation of these patients through metabolic stimulation, increased vascularization and oxygenation of directly affected tissues, effects of deep hyperthermia generated by the interaction of the current with the treated biological substrate, as well as the activation of tissue regeneration, the result of subthermal action. It is thus intended to improve signs such as global muscle capacity, which is essential for the recovery of the post-COVID-19 patients.

The hypothesis of this study is that current post-COVID-19 treatments can be significantly improved in order to prevent complications and ensure the patients' well-being.

DETAILED DESCRIPTION:
The new post-pandemic era has left sequelae in patients who presented the signs and symptoms of SARV-CoV2 and subsequently faced a positive for COVID-19. Such sequelae will be evident at various systemic levels of the affected patienta in the short, medium and long term future. One of these levels is musculoskeletal complications and injuries that have been documented throughout all scientific research since the beginning of massive infections worldwide.

SARS-CoV-2 is transmitted by penetrating the respiratory route (mostly), by fluid contact, and to a lesser extent, through the ocular pathway. In the field of neurology system, different forms of RF, nerve infiltrations, lymph node injuries, plantar fasciitis, spinal (peripheral) nerve disorders, etc. have been documented.

If the investigators focus on one of the most prevalent symptoms (those that affect the respiratory system), the bibliography that endorses that the RF could improve has been referenced.

The aim of this study is to assess the potential benefits of RF in patients with musculoskeletal problems which started after SARV-CoV-2 infection. The work proposed here aims to demonstrate the advantages of establishing RF as an excellent treatment for post-COVID-19 sequelae, due to its ability to reinforce immune action, modulate the inflammatory response and activate cellular and tissue regeneration.

The specific objectives of this research work are:

To demonstrate the efficacy of RF as a therapy in musculoskeletal pathologies derived from the sequelae of COVID-19.

To evidence and document the effects generated by the treatment with RF in the musculoskeletal system.

To estimate the level of benefit from RF in the musculoskeletal system treated and define the benefit/risk ratio.

To present and validate the therapy for the injuries under study that show significant improvements.

REGULATIONS

This clinical study will be carried out in accordance with the protocol, the principles established in the current revised version of the Declaration of Helsinki (Fortaleza, 2013) and in accordance with the applicable regulatory requirements.

The researcher is aware, when signing the protocol, of the obligation to adhere to the instructions and procedures described in it, and will ensure that the established provisions are strictly adhered to.

The study will not begin until the approval of the Research Ethics Committee has been obtained.

The principal investigator is responsible for ensuring that this protocol, the informed consent document, and any other information that is presented or facilitated to the possible subjects is reviewed and approved by the CEI. The Researcher agrees to allow direct access to the REC to all relevant documents.

INFORMED CONSENT.

In this case, patients must give their consent prior to being included in the study. The content and the procedure for obtaining it must be in accordance with all applicable legal requirements.

The investigator is responsible for obtaining the written informed consent of each patient participating in this study, after having explained in an understandable way, the nature, objectives, methods, expected benefits and possible risks of the study. The investigator must also explain to them that patients are completely free to refuse to participate in the study or to withdraw from it at any time, for whatever reason.

The study patients will give their consent, signing the corresponding model. For this purpose, each informed consent must be signed by both the investigator and the patient.

CONFIDENTIALITY.

All information related to the study is considered confidential in compliance with the confidentiality and custody of the data collected, in accordance with the 3/2018 Law on the protection of personal data (LOPDGDD), (article 5). Article 5.1 .f) of the RGPD states that personal data will be treated in such a way as to guarantee confidentiality and integrity In order to guarantee the confidentiality of the study data, only the main researcher and her team of collaborators will have access to it, the CEI and the pertinent health authorities.

FINANCING

The financing is assumed by the Gema León Physiotherapy and Rehabilitation Clinic. There is no direct economic consideration for this, although there is a dedication of time and work by the team of physiotherapists (social security, payroll, personal income tax, etc.) that is not economically remunerated and is assumed or absorbed this way. In addition, the RF technology (equipment and accessories) will be provided by the company INDIBA S.A., through a temporary assignment without any financial compensation either from the Gema León Physiotherapy Clinic, or from any patient. The treatment of these is completely free for them.

The patient must travel to the clinic facilities and it is the researcher who will be responsible for the treatment in it.

No difficulties are foreseen in its performance since it will be carried out using a schedule adapted to the patient that allows the study to be monitored.

It is intended to carry out a longitudinal study with the participation of 99 patients with elbow musculoskeletal pathology, who confirmed a positive test for COVID-19. The sample size for our study is large enough to detect a clinically important difference in the primary outcome (s). For this, the investigators reviewed references at the bibliographic level, in which paired studies obtained a statistically significant value, being able to support our study. If the sample size was insufficient but statistically significant, the investigators would resort to expanding the sample. The division of the sample is carried out at random within the established groups.

The patients will be divided into three groups: Group A or Placebo Group, which received the treatment with the machine turned off. Radiofrequency 448 Hz was administered to the affected area in two phases, depending on the electrode applied: 10 minutes of capacitive electrode and 35 minutes of resistive electrode, both with the machine turned off. Group B or Mixed Group, treatment with manual therapy and radiofrequency. Radiofrequency 448 Hz was administered to the affected area in two phases, depending on the electrode applied: 5 minutes of capacitive electrode and 25 minutes of resistive electrode. In addition, a specific joint physical therapy manual therapy treatment was also performed, in which pumping techniques were performed after the radiofrequency treatment.Group C or Manual Group, to which conventional manual therapy was applied for each case. Articulatory pumping techniques were applied towards the painful position with the aim of reducing it.

Thus we compare the therapies of groups A, B and C, of Musculoskeletal Pathologies.

All groups will be evaluated at the beginning, a second evaluation after 3 weeks and a third final control after 12 sessions. A fourth evaluation will be carried out after the last and final evaluation, 6 weeks after finishing the treatment. Each of the participants will be informed of the study, the objective, its possible benefits and the side effects that could arise. A) Therefore, each patient must give their free and confirmed consent through signature. Among the items in the methodology, the following stand out:

Primary data parameters: A series of questions will be asked to each of the patients about the conditions diagnosed during the disease and those suffered after the infection that are directly related to abnormalities to be assessed.

Secondary Data Parameters: The therapeutic protocol will be executed in the facilities of the Gema León Physiotherapy and Rehabilitation Clinic (Cordoba, Spain). Such RF therapeutic protocol will be implemented by application with an INDIBA® Activ device, whose function is to reduce inflammation, stimulate immunity and promote tissue regeneration. This will consist of a 30-minute treatment, composed by 5 minutes of treatment with the capacitive electrode and 25 minutes of the resistive electrode. A total of 12 sessions will be scheduled (two per week), and all processes will be documented from the beginning of therapy (the resources used will be provided by INDIBA and the Gema León Physiotherapy and Rehabilitation Clinic, whose supervision will be carried out by the direction of both).

Dependent Variables: variables of nominal type such as sex, age, vaccination, number of days with symptoms, type of symptom will be created. The patients will be grouped into 3 groups of 33 participants each (99 in total):

Placebo Group, which received the treatment with the machine turned off. Radiofrequency 448 Hz was administered to the affected area in two phases, depending on the electrode applied: 10 minutes of capacitive electrode and 35 minutes of resistive electrode, both with the machine turned off.

Experimental Mixed Group, treatment with manual therapy and radiofrequency. Radiofrequency 448 Hz was administered to the affected area in two phases, depending on the electrode applied: 5 minutes of capacitive electrode and 25 minutes of resistive electrode. In addition, a specific joint physical therapy manual therapy treatment was also performed, in which pumping techniques were performed after the radiofrequency treatment.

Convencional Manual Group, to which conventional manual therapy was applied for each case. Articulatory pumping techniques were applied towards the painful position with the aim of reducing it.

Independent Variables: In order to compare the variables between groups, different methods of pain threshold and function of the mentioned systems will be used, such as: Global Functionality Scale (GAF), Katz Index for Independence, Lawton and Brody Scale of Basic Activities, Barthel index for disability, European Quality of Life 5-D Questionnaire (EURO- QoL 5-D) for quality of life, Tinetti test for gait and balance, joint amplitude scale measured with the goniometer (goniometry), strength muscle dynamometer (Dynamometry), pain index (Visual Analogue Scale (VAS), reflectivity measurement with the Wartenberg Scale for bone tendon reflexes (ROTs), examination of sensitivity from evaluation of dermatomes. The statistical analysis is based on variables of nominal type mostly, which are suitable for the Chi square test with a significance value of 95% for the results (p <0.05). However, if there are numerical data that must be compared between groups, the analysis will be used for ANOVA test with the same significance value for the comparison between results.

ELIGIBILITY:
Inclusion Criteria:

* Patients between the ages of 18 and 60.
* Patients with a positive diagnosis of COVID-19.
* Patients with post-COVID-19 sequelae with elbow musculoskeletal diseases.
* Patients who signed the informed consent.

Exclusion Criteria:

* Patients aged before 18 years and after 60 years.
* Healthy people with no history of elbow musculoskeletal diseases
* Patients with secondary diseases that could directly affect the systems to be evaluated who were not diagnosed positive for COVID-19.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 99 (Actual)
Dates: Start 2021-06-16 (Actual); Primary Completion 2022-06-21 (Actual); Study Completion 2022-07-20 (Actual)

PRIMARY OUTCOMES:
Joint range of motion was measured | 3 months
  Measurements were taken using a goniometer of at least two joint movement axes in each casMeasurements were taken using a goniometer of at least two joint movement axes in each case
A muscle assessment was performed. | 3 months
  Strength measurements were taken using a dynamometer. The peak torque during a 5-second concentric contraction was measured. This contraction was repeated a total of three times, with the average of the three measurements taken as the final result.

SECONDARY OUTCOMES:
Upper Limb Functional Index questionnaire | 3 months
  A total of 20 questions with responses ranging from 0 to 4. Optimal total score: 80. Minimum score: 0. Maximum score: 80.
Lower Extremity Functional Scale for the lower limb. | 3 months
  25 questions with responses ranging from 0 to 4. Optimal total score: 100. Minimum score: 0. Maximum score: 100.
Visual Analogue Scale for pain (VAS) | 3 months
  which allows for the classification of the patient's pain on a scale from 0 (no pain) to 10 (unbearable pain)
Patient independence (Katz Index) | 3 months
  Questions about activities of daily living were provided. Minimum value: 0 (ability to perform basic activities of daily living). Maximum value: 1 (inability to perform basic activities of daily living). Optimal value: 0.

OTHER OUTCOMES:
Relevant data such as the duration of each patient's symptoms | 3 months
  Whether they had been previously vaccinated or not

CONTACTS AND LOCATIONS:
Overall Officials: Gema Leon Bravo, Principal Investigator — Departamento de Enfermería, Farmacología y Fisioterapia de la Universidad de Córdoba
Locations (1):
- Gema León Physiotherapy and Rehabilitation Clinic, Córdoba, Andalusia, Spain

IPD SHARING:
Plan to Share IPD: No
The request for the data will be studied and considered upon prior and justified request.

REFERENCES:
- [Background] Bito T, Tashiro Y, Suzuki Y, Kajiwara Y, Zeidan H, Kawagoe M, Sonoda T, Nakayama Y, Yokota Y, Shimoura K, Tatsumi M, Nakai K, Nishida Y, Yoshimi S, Tsuboyama T, Aoyama T. Acute effects of capacitive and resistive electric transfer (CRet) on the Achilles tendon. Electromagn Biol Med. 2019;38(1):48-54. doi: 10.1080/15368378.2019.1567525. Epub 2019 Jan 19. PMID 30663425
- [Background] Tashiro Y, Hasegawa S, Yokota Y, Nishiguchi S, Fukutani N, Shirooka H, Tasaka S, Matsushita T, Matsubara K, Nakayama Y, Sonoda T, Tsuboyama T, Aoyama T. Effect of Capacitive and Resistive electric transfer on haemoglobin saturation and tissue temperature. Int J Hyperthermia. 2017 Sep;33(6):696-702. doi: 10.1080/02656736.2017.1289252. Epub 2017 Feb 19. PMID 28139939
- [Background] Arena M. Radiofrequency A 448 kHz in the treatment of muscle spasticity in a dog with C2-C3 spinal cord injury. 2018. 12-3.
- [Background] Erdine S, Ozyalcin NS, Cimen A, Celik M, Talu GK, Disci R. Comparison of pulsed radiofrequency with conventional radiofrequency in the treatment of idiopathic trigeminal neuralgia. Eur J Pain. 2007 Apr;11(3):309-13. doi: 10.1016/j.ejpain.2006.04.001. Epub 2006 Jun 9. PMID 16762570
- [Background] Pérez-Cajaraville J., Aseguinolaza Pagola M., Molina Tresaco P., Arranz Duran J., Abejon Gonzalez D.. Trigeminal neuralgia: Gasser ganglion radiofrecuency. Rev. Soc. Esp. Dolor [Internet]. 2013 Apr [cited 2025 July 16] ; 20( 2 ): 89-100. Available from: http://scielo.isciii.es/scielo.php?script=sci_arttext&pid=S1134-80462013000200007&lng=en. https://dx.doi.org/10.4321/S1134-80462013000200007.
- [Background] Martínez Rubio A, Bordas JR. Treatment of asthma by capacitive electrical transfer (ECT). Rehab Fis. 1992; 3 (13): 18-9.
- [Background] Alves A, Quispe A, Ávila A, Valdivia A, Chino J, Vera O. Brief history and pathophysiology of COVID-19. Diagnostic Guide and COVID-19 Treatment in Ter Intensive Units for Boliv [Internet]. 2020; 61 (1): 77-86.
- [Result] Bito T, Suzuki Y, Kajiwara Y, Zeidan H, Harada K, Shimoura K, Tatsumi M, Nakai K, Nishida Y, Yoshimi S, Kawabe R, Yokota J, Yamashiro C, Tsuboyama T, Aoyama T. Effects of deep thermotherapy on chest wall mobility of healthy elderly women. Electromagn Biol Med. 2020 Apr 2;39(2):123-128. doi: 10.1080/15368378.2020.1737803. Epub 2020 Mar 4. PMID 32131642